CLINICAL TRIAL: NCT04369261
Title: A Multicenter, Prospective Observational Study to Evaluate the Injection Site Reactions of Synovian® Inj. in Patients With Osteoarthritis in the Knee
Brief Title: Observational Study of Synovian® Inj. in Patients With Osteoarthritis in the Knee
Status: Completed | Type: Observational
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-HAOS006
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis in the Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Synovian® — Synovian® Inj.

SUMMARY:
This is an observational study to evaluate the injection site reactions of Synovian® Inj. in patients with osteoarthritis in the knee

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patient of over 19 years of age
* A patient diagnosed with knee osteoarthritis
* A patient who has been informed of the purpose, method of the study and signed the written informed consent form.

Exclusion Criteria:

* A patient who shows hypersensitive reaction to the Synovian® Inj. or to the ingredients of Synovian® Inj.
* A patient with infection at the joint
* A patient with skin infection or skin disease at the injection area
* A patient diagnosed with osteoarthritis with the Kellgren & Lawrence Grade IV in X-ray within 12 months before enrollment of this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient from hospital and clinic as well
Sampling Method: Probability Sample
Enrollment: 1949 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
safety endpoints | Week 2
  injection site reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University GURI Hospital, Guri-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
not decided

REFERENCES:
- [Derived] Jang KM, Park YG, Choi WK, Chung YY, Kim KK, Lee JW, Lee SJ, Eom Y, Yang JH. Safety of a single intra-articular injection of LBSA0103 hyaluronic acid in patients with osteoarthritis of the knee: a multicenter, single-arm, prospective, cohort study. Curr Med Res Opin. 2021 Sep;37(9):1573-1580. doi: 10.1080/03007995.2021.1950132. Epub 2021 Jul 15. PMID 34192989